CLINICAL TRIAL: NCT05100745
Title: A Non-significant Risk Clinical Study to Assess Changes in Perfusion Resulting From Application of the VibratoSleeve, a Therapeutic Ultrasound (TUS) Phased Array, for Patients With Peripheral Arterial Disease (PAD)
Brief Title: A Non-significant Risk Clinical Study to Assess Perfusion Changes With Application of a TUS for Patients With PAD
Acronym: Concerto
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vibrato Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 21-001
Record Dates: First submitted 2021-10-21; First posted 2021-10-29 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Peripheral Arterial Disease
Keywords: Therapeutic Ultrasound (TUS); Peripheral Artery Disease (PAD); Critical Limb Ischemia (CLI)
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Intervention Model Description: Prospective, double-blinded, randomized controlled trial to evaluate the feasibility of TUS in the treatment of PAD.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Clinicians and subjects in both the active and sham group will be blinded to the randomized treatment assignments until 2-month follow-up visit. The sham and active devices will appear the same and appear to be utilized in the same manner. Only the Vibrato Medical person controlling the treatment device will be aware of the respective randomization for each subject. The second phase of this study, crossing over from sham to active treatment will not be concealed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Activated Therapy (Experimental): Therapy: these subjects will undergo 30 treatments with an activated Vibratosleeve TUS device.
  Interventions: Device: Therapeutic Device
- Sham Therapy (Sham Comparator): An inactive (sham) device will be used in these subjects for the first 30 treatments followed by a 30-treatment regimen with an activated VibratoSleeve TUS device after crossover.
  Interventions: Device: Therapeutic Device

INTERVENTIONS:
Device: Therapeutic Device — This device delivers ultrasound energy to the targeted area of the lower limb.
  Other Names: VibratoSleeve TUS Device

SUMMARY:
The objective of the clinical trial is to gather evidence on the safety, performance and clinical efficacy Vibrato Sleeve TUS in people with peripheral artery disease (PAD).

DETAILED DESCRIPTION:
Subjects will be randomized to a test or control group and will receive an active or sham Vibrato Sleeve respectively.

Those randomized to the control arm will undergo therapy sessions with a sham Vibrato Sleeve device and two months of follow-up. Upon completion of the 2-month follow-up visit, subjects will be informed of their randomization assignment. Subjects in the sham arm will be allowed to crossover to a treatment regimen that uses an active Vibrato Sleeve device and will follow the same visit schedule as the active test group.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥22.
2. Diagnosis of infrapopliteal PAD.
3. Rutherford class 4 or 5 as determined by the investigator.
4. Toe Brachial Index (TBI) ≤ 0.6 OR Toe Blood Pressure ≤ 50 mmHg.

Exclusion Criteria:

1. Prior stenting in posterior tibial, anterior tibial or peroneal artery.
2. Re-vascularization procedure within 25 days prior to enrollment in the study. (Note: Patients who had re-vascularization procedure earlier than 25 days prior to enrollment are eligible for enrollment if they meet other criteria).
3. Ulcers, cellulitis, or skin breakdown in treatment areas (posterior calf).
4. History or diagnosis of severe chronic venous insufficiency or mixed arterio-venous disease.
5. Acute limb ischemia within 30 days prior to treatment.
6. History or diagnosis of deep venous thrombosis below the knee in treatment leg.
7. Uncontrolled diabetes defined as HbA1c greater than 10%.
8. Ongoing hyperbaric oxygen treatment (HBOT)
9. Any conditions that, in the opinion of the investigator, may render the patient unable to complete the study or lead to difficulties for patient compliance with study requirements, or could confound study data.

9. Patient's enrollment in another investigational study that has not completed the required primary endpoint follow-up period (Note: Patients involved in a long-term surveillance phase of another study are eligible for enrollment in this study).

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Changes in foot perfusion | 4 months
  Mean difference between pre-treatment (baseline) and/or last sham treatment with post-treatment measurements, including the 2-month follow-up.

SECONDARY OUTCOMES:
Adverse Events | up to and including the 2-month follow-up visit for test and control subjects.
  Analysis of all reported device-related adverse events throughout each subject's participation.
Subject Questionnaire | up to and including the 2-month follow-up visit for test and control subjects.
  Questions will be based on each treatment session and what each subject felt and observed.

CONTACTS AND LOCATIONS:
Locations (1):
- Vascular & Interventional Specialists of Orange County, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No
Data summaries, group outcomes, and study conclusions will be shared with other researchers. Individual participant data will not be shared.

REFERENCES:
- [Result] Nazer B, Ghahghaie F, Kashima R, Khokhlova T, Perez C, Crum L, Matula T, Hata A. Therapeutic Ultrasound Promotes Reperfusion and Angiogenesis in a Rat Model of Peripheral Arterial Disease. Circ J. 2015;79(9):2043-9. doi: 10.1253/circj.CJ-15-0366. Epub 2015 Jun 9. PMID 26062950